CLINICAL TRIAL: NCT05158465
Title: Project Motivate Me Clinical Trial: Oral Hygiene Intervention for Adolescents
Brief Title: Oral Hygiene Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Vista Community Clinic (Unknown)
Responsible Party: Principal Investigator, Tracy L Finlayson, Principal Investigator, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2021-0276
Record Dates: First submitted 2021-06-19; First posted 2021-12-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Intervention and control groups will be enrolled and followed over one-month.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing and Assessments (Experimental): Two 1 hour assessments. At each assessment, participant will complete a survey, supply a saliva sample, do a toothpick test, and take a plaque photo. Three one-on-one, half hour educational and skill-building MI sessions will address: proper oral hygiene technique, bacteria and dental caries process, and nutrition. Intervention group adolescents will also receive three calls over one month reinforcing their hygiene behavior goals.
  Interventions: Behavioral: Motivational Interviewing
- Assessments Only (No Intervention): Two 1 hour assessments. At each assessment, participant will complete a survey, supply a saliva sample, do a toothpick test, and take a plaque photo.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Intervention will include 3 one-on-one motivational interviewing sessions and 3 follow-up calls with a trained MI health educator. These sessions aim to promote better oral hygiene and oral health.
  Arms: Motivational Interviewing and Assessments

SUMMARY:
The purpose of this study is to promote oral hygiene behaviors (toothbrushing, flossing) and oral health with high-risk adolescents in San Diego, CA, through a Motivational Interviewing (MI) Intervention.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will evaluate the efficacy of a new, brief motivational interviewing (MI)- based intervention and assess its impact on several sets of outcomes among 14-19 years old Latino adolescents: clinical oral health and hygiene indices, counts of biological caries-causing bacteria, and oral hygiene behaviors. Three one-on-one, half hour educational and skill-building MI sessions will address: proper oral hygiene technique, bacteria and dental caries process, and nutrition. Intervention group adolescents will also receive three telephone calls (one/month reinforcing their hygiene behavior goals. Outcomes will be assessed at baseline (T1), and at one-month (T2), after the intervention group received three MI sessions and three booster calls.

Aim 1. To develop and assess a new Motivational Interviewing (MI)-based behavioral oral health intervention for Latino adolescents in a randomized controlled trial (RCT) design. Finalize all intervention educational materials and scripts and assessment tools.

Aim 2. To assess the efficacy of the brief intervention on reductions in clinically determined outcomes among intervention versus control participants.

Aim 3. To assess the efficacy of the brief intervention on reductions in the presence and count of two types of biological bacteria involved in the dental caries disease process.

Aim 4. To assess the efficacy of the brief intervention in increasing the frequency of daily oral hygiene behaviors, including properly brushing, flossing, and rinsing.

Aim 5. Conduct process evaluation via two focus groups post-intervention to assess the acceptability and feasibility of the intervention and assessments (one for intervention group; one for control group).

The investigators hypothesize that the intervention group will see improved clinical outcomes, lower bacteria counts, and better oral hygiene behavior than the control group.

ELIGIBILITY:
Inclusion Criteria:

* self identifies as Mexican or Mexican-American
* living in Northern San Diego County
* speaks English
* able to access stable internet
* participates in 1 or more program or service at VCC

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Plaque Score at 1 month | At baseline and post-intervention (after about one month)
  Plaque levels will be scored for each participant based on photographs taken after the use of a plaque disclosure tablet. This will be scored as low (minimum), moderate, or high (maximum). Lower is better.
Change from Baseline in Gum Bleeding at 1 month. | at baseline, and post-intervention (after about one month)
  Each participant will use a toothpick to probe 14 points in the mouth (7 points in the maxillary anterior teeth and 7 points in the mandibular anterior teeth). At each point, if the participant bleeds, they are given a score of "1". Then the score is added up at the end of probing each point. Minimum score is 1 and maximum score is 14. Lower score is better and higher score is worse.
Change from Baseline Weekly Toothbrushing at 1 month. | at baseline, and post-intervention (after about one month)
  Each participant will self-report frequency of toothbrushing in the past 7 days on a survey. This will be scored as a continuous count (minimum is zero, no set maximum) and whether or not they met ADA recommended guidelines for twice daily brushing. Higher frequency is better.
Change from Baseline in Weekly Flossing at 1 month. | at baseline, and post-intervention (after about one month)
  Each participant will self-report frequency of flossing in the last 7 days on a survey. This will be scored as a continuous count (minimum is zero, no set maximum) and whether or not they met ADA recommended guidelines for once daily flossing. Higher frequency is better.
Change from Baseline in Weekly Rinsing at 1 month. | at baseline, and post-intervention (after about one month)
  Each participant will self-report frequency of rinsing with water in the last 7 days on a survey. This will be scored as a continuous count (minimum is zero, no set maximum). Higher frequency is better.
Change from Baseline Oral Hygiene at 1 month. | at baseline, and post-intervention (after about one month)
  Each participant's oral hygiene skill level will be assessed and scored as poor (minimum), fair, good, or excellent (maximum) based on execution of specific micro-behaviors for brushing and flossing. Higher is better.
Change from Baseline Count in S. Mutans Bacteria in Saliva at 1 month. | at baseline, and post-intervention (after about one month)
  Saliva samples will be collected using Zymo collection kits to run qPCR analysis, which will yield information on whether or not bacteria is present (yes/no), and relative and absolute counts of S. mutans bacteria. Minimum is zero, no set maximum. Lower is better.
Change from Baseline Count in S. sobrinus Bacteria in Saliva at 1 month. | at baseline, and post-intervention (after about one month)
  Saliva samples will be collected using Zymo collection kits to run qPCR analysis, which will yield information on whether or not bacteria is present (yes/no), and relative and absolute counts of S. sobrinus bacteria. Minimum is zero, no set maximum. Lower is better.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Finlayson, PhD, Principal Investigator — San Diego State University
Locations (1):
- Vista Community Clinic, Vista, California, United States

IPD SHARING:
Plan to Share IPD: No